CLINICAL TRIAL: NCT01161680
Title: A Prospective Baseline Assessment of the Risk of Osteoporosis in Patients With Chronic Obstructive Lung Disease and Outcomes After 2 Years; a Pilot Study
Brief Title: Breathing and Bones Initiative
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Mark Fitzgerald, Principal Investigator, University of British Columbia
Other Study IDs: H10-00983
Record Dates: First submitted 2010-06-22; First posted 2010-07-13 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Osteoporosis; Obstructive Lung Disease
Keywords: Cross sectional and Longitudinal Observational study
MeSH Terms: conditions — Osteoporosis; Lung Diseases, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This project will examine the current diagnosis and treatment of bone health in patients with obstructive airway disease. Patients will be referred to The Osteoporosis Centre of BC (OCBC) by their respirologist to be assessed for osteoporosis including Dual Energy Xray Absorptiometry (DXA) scan. Previous chest xrays and will be accessed and examined for vertebral fractures, diagnostic of osteoporosis. The lung and bone data will be entered into a database. This will allow us to explore the relationship of lung disease parameters to osteoporosis predictors, eventually determining a respirology patient population who are at high risk of fracture. Longitudinal evaluation of bone health and its relationship to respiratory parameters over time will be explored by follow-up evaluations at 12 and 24 months.

DETAILED DESCRIPTION:
Research Method:

1. Selected respirologists' practices will identify patients at risk of osteoporosis (according to Osteoporosis Canada Guidelines):

   1. Who have not had a bone density test in the past 2 years and
   2. Who are not already taking osteoporosis pharmacotherapy.
   3. Other patients not meeting these criteria can also be referred at the discretion of the physician
2. Patients will be given a choice on whether they wish to be referred to the Osteoporosis Centre of BC (Vancouver) through an expedited simple referral system OR they may have their information sent to their referring/family doctor discussing the need for referral for an evaluation of bone health and follow up

   i. Informed consent obtained with an Ethics Committee approved Informed Consent Form. Informed consent will be obtained from all patients who will be followed by the research team. The consent will allow the researchers to use clinical data and imaging for observational research; participation in the research will be optional and will not affect patient ability to obtain information on their bone health at OCBC.

ii. A standard, full evaluation will be undertaken on a single visit (DXA bone densitometry, consultation with endocrinologist or geriatrician). Screening for secondary causes of osteoporosis including Vitamin D status through blood tests will occur at a community laboratory. All information obtained from these tests being reviewed by the physicians and clinical treatment decisions will be made based on standard practice.

iii. Densitometry with OCBC research-calibrated DXA will permit meaningful clinical follow-up .

Respirologists' office process:

1. Men and women over age 65 with obstructive airways disease would be asked if they have had a bone density test in the past 2 years and if they are currently taking an osteoporosis therapy (alendronate, risedronate, zoledronate, etidronate, , raloxifene, calcitonin, estrogen)

2 If the answer is no, the respirologists would

Explain standard of care for patients at risk of osteoporosis and then

1. Recommend to the referring physician that an osteoporosis evaluation be conducted (non-study) or
2. Ask the patient if they would be interested in taking part of the observational study. If patient wishes to participate a consent form would be given to the subject and the patient would be asked for permission to have the research coordinator call them in 2-3 days to discuss the study. The respirologist would then generate an expedited referral to the Osteoporosis Centre of BC (candidate for observational study).

The research coordinator would contact the subject by telephone and with scripted call speak to the subject and answer any questions pertaining to the study. During this call the research coordinator would determine whether the subject would like to meet prior to the appointment so that informed consent could be obtained. Informed consent would be obtained at the OCBC prior to the patient's appointment. If the patient does not wish to consent to the study but is referred clinically, they will not meet with the study coordinator, but they will still be able to access all usual clinical services provided by OCBC.

i. A simple one-page referral faxed to Osteoporosis Centre of BC

ii. All arrangements made either with respirologists' office or directly with the patient by OCBC

iii. Consultation reports sent back to both the referring doctor (respirology) and family doctor

Data from osteoporosis clinical history, fracture history, medication history, chemistries, and DXA will be collected with data on respiratory function. A database would be made for later analysis and correlation.

Chest Xray films taken in the last 2 years would be reviewed. Chest CT or other imaging will be evaluated for vertebral compression fractures (a very potent risk factor for future fragility fracture).

Statistical Analysis:

This study is observational and descriptive data will be produced. Regressions of continuous variables will be analyzed using Pearson correlation coefficients and parametric variables analyzed by Chi Squared testing.

ELIGIBILITY:
Inclusion Criteria:

* men and women over 65 years of age with obstructive airway disease being seen by a respirologist in their clinical practices

Exclusion Criteria:

* less than 65 years of age
* patient has had bone density scan within the last 2 years
* patient is currently being treated for osteoporosis (alendronate, risedronate, zoledronate, etidronate, clodronate, raloxifene, calcitonin, estrogen)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients will be drawn from specified respirology clinics: The Lung Centre (VCH) and The Pacific Lung Centre (PHC)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-07; Primary Completion 2011-09 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To determine the prevalence of osteoporosis in the respiratory disease population, as determined by bone density and fragility fracture.

SECONDARY OUTCOMES:
To associate osteoporosis with severity of pulmonary disease in respirology disease patients.

CONTACTS AND LOCATIONS:
Overall Officials: Mark FitzGerald, MD, Principal Investigator — University of British Columbia
Locations (3):
- Canada (3):
  - The Osteoporosis Centre of BC (Bone Consultaton and Bone Mineral Density), Vancouver, British Columbia
  - The Lung Centre, Vancouver Coastal Health, 7th Floor 2775 Laurel Street, Vancouver, British Columbia
  - The Pacific Lung Centre, Providence Health Care, Vancouver, British Columbia

REFERENCES:
- [Background] Yende S, Waterer GW, Tolley EA, Newman AB, Bauer DC, Taaffe DR, Jensen R, Crapo R, Rubin S, Nevitt M, Simonsick EM, Satterfield S, Harris T, Kritchevsky SB. Inflammatory markers are associated with ventilatory limitation and muscle dysfunction in obstructive lung disease in well functioning elderly subjects. Thorax. 2006 Jan;61(1):10-6. doi: 10.1136/thx.2004.034181. Epub 2005 Nov 11. PMID 16284220
- [Background] Kjensli A, Mowinckel P, Ryg MS, Falch JA. Low bone mineral density is related to severity of chronic obstructive pulmonary disease. Bone. 2007 Feb;40(2):493-7. doi: 10.1016/j.bone.2006.09.005. Epub 2006 Oct 13. PMID 17049326
- [Background] Watz H, Waschki B, Boehme C, Claussen M, Meyer T, Magnussen H. Extrapulmonary effects of chronic obstructive pulmonary disease on physical activity: a cross-sectional study. Am J Respir Crit Care Med. 2008 Apr 1;177(7):743-51. doi: 10.1164/rccm.200707-1011OC. Epub 2007 Nov 29. PMID 18048807
- [Background] Donaldson GC, Seemungal TA, Patel IS, Bhowmik A, Wilkinson TM, Hurst JR, Maccallum PK, Wedzicha JA. Airway and systemic inflammation and decline in lung function in patients with COPD. Chest. 2005 Oct;128(4):1995-2004. doi: 10.1378/chest.128.4.1995. PMID 16236847
- [Background] Jorgensen NR, Schwarz P, Holme I, Henriksen BM, Petersen LJ, Backer V. The prevalence of osteoporosis in patients with chronic obstructive pulmonary disease: a cross sectional study. Respir Med. 2007 Jan;101(1):177-85. doi: 10.1016/j.rmed.2006.03.029. Epub 2006 May 4. PMID 16677808
- [Background] Maggi S, Siviero P, Gonnelli S, Schiraldi C, Malavolta N, Nuti R, Crepaldi G; EOLO Study Group. Osteoporosis risk in patients with chronic obstructive pulmonary disease: the EOLO study. J Clin Densitom. 2009 Jul-Sep;12(3):345-52. doi: 10.1016/j.jocd.2009.05.003. PMID 19647671
- [Background] Blake GM, Fogelman I. The clinical role of dual energy X-ray absorptiometry. Eur J Radiol. 2009 Sep;71(3):406-14. doi: 10.1016/j.ejrad.2008.04.062. Epub 2009 Aug 3. PMID 19647962
- [Background] Papaioannou A, Parkinson W, Ferko N, Probyn L, Ioannidis G, Jurriaans E, Cox G, Cook RJ, Kumbhare D, Adachi JD. Prevalence of vertebral fractures among patients with chronic obstructive pulmonary disease in Canada. Osteoporos Int. 2003 Nov;14(11):913-7. doi: 10.1007/s00198-003-1449-5. Epub 2003 Oct 9. PMID 14551675
- [Background] Wanner A, Chediak AD, Csete ME. Airway mucosal blood flow: response to autonomic and inflammatory stimuli. Eur Respir J Suppl. 1990 Dec;12:618s-623s. PMID 1981675
- [Background] Leech JA, Dulberg C, Kellie S, Pattee L, Gay J. Relationship of lung function to severity of osteoporosis in women. Am Rev Respir Dis. 1990 Jan;141(1):68-71. doi: 10.1164/ajrccm/141.1.68. PMID 2297189
- [Background] Rossi C, Chianchiano N, Bertolino G, Perino A, Cittadini E. Ultrasonography and blood flow velocity waveform assessment in human fetuses. Acta Eur Fertil. 1991 May-Jun;22(3):147-9. PMID 1803824
- [Background] Anderson D, Macnee W. Targeted treatment in COPD: a multi-system approach for a multi-system disease. Int J Chron Obstruct Pulmon Dis. 2009;4:321-35. doi: 10.2147/copd.s2999. Epub 2009 Sep 1. PMID 19750192
- [Background] Walsh LJ, Lewis SA, Wong CA, Cooper S, Oborne J, Cawte SA, Harrison T, Green DJ, Pringle M, Hubbard R, Tattersfield AE. The impact of oral corticosteroid use on bone mineral density and vertebral fracture. Am J Respir Crit Care Med. 2002 Sep 1;166(5):691-5. doi: 10.1164/rccm.2110047. PMID 12204867
- [Background] McEvoy CE, Ensrud KE, Bender E, Genant HK, Yu W, Griffith JM, Niewoehner DE. Association between corticosteroid use and vertebral fractures in older men with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1998 Mar;157(3 Pt 1):704-9. doi: 10.1164/ajrccm.157.3.9703080. PMID 9517579
- [Background] Bolton CE, Ionescu AA, Shiels KM, Pettit RJ, Edwards PH, Stone MD, Nixon LS, Evans WD, Griffiths TL, Shale DJ. Associated loss of fat-free mass and bone mineral density in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2004 Dec 15;170(12):1286-93. doi: 10.1164/rccm.200406-754OC. Epub 2004 Sep 16. PMID 15374843
- [Background] Vestergaard P, Rejnmark L, Mosekilde L. Fracture risk in patients with chronic lung diseases treated with bronchodilator drugs and inhaled and oral corticosteroids. Chest. 2007 Nov;132(5):1599-607. doi: 10.1378/chest.07-1092. Epub 2007 Sep 21. PMID 17890464
- [Background] Ferguson GT, Calverley PMA, Anderson JA, Jenkins CR, Jones PW, Willits LR, Yates JC, Vestbo J, Celli B. Prevalence and progression of osteoporosis in patients with COPD: results from the TOwards a Revolution in COPD Health study. Chest. 2009 Dec;136(6):1456-1465. doi: 10.1378/chest.08-3016. Epub 2009 Jul 6. PMID 19581353
- [Background] Madsen H, Brixen K, Hallas J. Screening, prevention and treatment of osteoporosis in patients with chronic obstructive pulmonary disease - a population-based database study. Clin Respir J. 2010 Jan;4(1):22-9. doi: 10.1111/j.1752-699X.2009.00138.x. PMID 20298414
- [Background] Brown JP, Josse RG; Scientific Advisory Council of the Osteoporosis Society of Canada. 2002 clinical practice guidelines for the diagnosis and management of osteoporosis in Canada. CMAJ. 2002 Nov 12;167(10 Suppl):S1-34. PMID 12427685